CLINICAL TRIAL: NCT07209358
Title: A Multi-Centre, Observer-Blinded, Randomized Controlled Trial of EDX110 for the Treatment of Diabetic Foot Ulcers
Brief Title: EDX110 Randomized Control Trial for Treatment of DFUs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WC-24-447
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Wound Heal; Diabetic Foot Ulcer
Keywords: Hard to heal wounds
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Observer blinded assessment of wound closure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EDX110 with Standard of Care (SOC) (Active Comparator): Diabetic Foot Ulcer (DFU) DFU treatment with EDX110 wound dressing and SOC
  Interventions: Device: EDX110
- Standard of Care (SOC) (No Intervention): Diabetic Foot Ulcer (DFU) DFU treatment with using only traditional Standard of Care (SOC)

INTERVENTIONS:
Device: EDX110 — EDX110 wound dressing system EDX110 is a dressing system comprising two layers that allows the generation of nitric oxide (NO) in situ, enables adequate moisture management and facilitates debridement
  Arms: EDX110 with Standard of Care (SOC)

SUMMARY:
Prospective, multi-centered, observer blinded, pre-market study, 1:1 randomized control trial, to determine if addition of EDX110 dressing system to standard of care leads to an improvement in diabetic foot ulcers healing compared to just using standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Participants at least 18 years old and willing to participate in all procedures and follow-up evaluations necessary to complete the study.
* The participant must have an index ulcer meeting the following characteristics:

  1. Non-healing DFU defined as; at least 4 weeks prior to enrolment the ulcer has failed to progress on a healing trajectory.
  2. Full-thickness wound; defined as Wagner Diabetic Foot Ulcer Grade 1 - superficial ulcer of skin or subcutaneous tissue.
  3. Located on the anatomical foot; defined as distal to the medial or lateral malleolus.
* Presents with or without clinical signs of superficial infection. Infection is defined using International Working Group of the Diabetic Foot (IWGDF) PEDIS classification and for the purpose of inclusion infections must be PEDIS grade 1 (Mild); Infected: At least two of these items are present: Local swelling or induration Erythema >0.5 but <2 cm2 around the wound, Local tenderness or pain, Local increased warmth, Purulent discharge.
* Ulcer duration at randomization must be present for ≥1 month but less than <24 months in duration.
* Post-debridement wound area is ≥0.1 cm2 and ≤25 cm2.
* If two or more ulcers either mono or bilateral are present, the index ulcer must additionally be:

  1. The ulcer with the largest wound area, as long as it meets all other criteria.
  2. ≥3cm distance from any other ulcer on the affected limb
* Known history of type 1 or type 2 diabetes (confirmed by the subject's medical history).
* HgbA1c <12% (NGSP) OR 108 mmol/mol (IFCC) OR average blood glucose 298 mg/DL.
* Participant has adequate circulation to the affected extremity as defined by Wound, Ischemia, foot Infection (WIfI) Ischemia grades 0-1 (no PAD to Mild PAD).
* Participants are required to have either.

  1. Ankle-Brachial Index (ABI) by Doppler: ≥0.6 OR Toe-Brachial Index (TBI) ≥ 0.5
  2. OR Dorsum transcutaneous oxygen test (TcPO2): >40 mm/Hg

Exclusion Criteria:

* Participants with wounds that have any of the following characteristics:

  1. Wagner Grade 2 - ulcers extend into tendon, bone, or capsule
  2. Grade 3 - deep ulcer with osteomyelitis, or abscess
  3. Grade 4 - partial foot gangrene
  4. Grade 5 - whole foot gangrene
* Infections that are classified as:

  1. PEDIS 3 (Moderate): Infection with no systemic manifestations and involving: Erythema extending ≥2 cm2 from the wound margin, and/or tissue deeper than skin and subcutaneous tissues (e.g., tendon, muscle, joint, and bone).
  2. PEDIS 4 (Severe): All of the above in PEDIS 3 plus manifestations (of the systemic inflammatory response syndrome [SIRS]).
  3. In addition, any diabetic foot infections with; Confirmed underlying bone involvement (osteomyelitis) based on; imaging (plain X-ray, CT or MRI), clinical examination (exposed bone or positive probe to bone test) or culture/histopathology of a bone specimen
  4. OR Cellulitis/lymphangitis/soft tissue gas or necrotizing fasciitis originating from the wound site.
* Tunnelling, Cavity or undermining wounds.
* Known or suspected local skin malignancy at the site of the ulcer.
* A wound that is actively bleeding. This does not exclude enrollment once active bleeding has stopped (hemostasis).
* Gross Foot deformities that would interfere with proper off-loading or proper wound healing i.e. non-active charcot foot, rocker bottom foot, gross digital deformities.
* Active Charcot deformity.
* Wound duration >2 years.
* Participants receiving any of the following prior therapies. In the last 30 days:

  1. Has required systemic corticosteroids >10mg/kg/day OR
  2. Participant has required Chemoradiation (chemotherapy and/or radiation therapy) to treat cancer and is immunocompromised OR
  3. Participant is anticipated to require such medications during the study period.
  4. Study ulcer treatment with any advanced therapy, including, biomedical or topical growth factors, tissue engineered materials (e.g., Apligraf or Dermagraft), sterilized placental allografts (EpiFix, NovaFix, etc.), or other scaffold materials (e.g., OASIS® Wound Matrix, MatriStem Wound Matrix).
  5. Has undergone any amputation to the affected leg.
* Known hypersensitivity to constituents of the product.
* Presence of any condition (including current drug or alcohol abuse, medical or psychiatric condition) that is likely to impair understanding of, or compliance with the study protocol in the judgement of the Investigator.
* Women of childbearing age (women aged <55 years who have not undergone menopause) who are:

  1. Pregnant at time of enrolment
  2. Breast-feeding
* Concurrent enrolment in any other study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound Closure | 16 Weeks
  Incidence of complete wound closure at 16 weeks in participants with DFU who are receiving standard of care (SOC) versus participants receiving EDX110 and SOC. Wound closure is defined as 100% reepithelialization of the wound without drainage.

SECONDARY OUTCOMES:
Time to Wound Closure | 16 Weeks
  Time to complete wound closure during treatment period in participants with DFU who are receiving standard of care (SOC) versus participants receiving EDX110 and SOC.
Percent Area Reduction 4 weeks | 4 Weeks
  The difference in the mean Percent Area of Reduction (PAR) at 4 weeks compared to baseline in participants with DFU who are receiving standard of care (SOC) versus participants receiving EDX110 and SOC.
Percent Area Reduction 16 weeks | 16 weeks
  The difference in the mean Percent Area of Reduction (PAR) at 16 weeks compared to baseline in participants with DFU who are receiving standard of care (SOC) versus participants receiving EDX110 and SOC.
Wound closure at 24 weeks | 24 weeks
  Incidence of complete wound closure at 24 weeks in participants with DFU who are receiving standard of care (SOC) versus participants receiving EDX110 and SOC. Wound closure is defined as 100% reepithelialization of the wound without drainage.

OTHER OUTCOMES:
Hospitalizations relating to the target ulcer | 16 Weeks
  Determine if the use of EDX110 leads to a reduction of the patient being hospitalized due to adverse events or complications related to their target ulcer.
Amputations relating to the target ulcer | 16 Weeks
  Determine if use of EDX110 leads to reduction in the occurrences of an amputation of the leg, foot, or toes due to the target ulcer.
Systemic antibiotic usage during the 16-week treatment period | 16 Weeks
  Determine if the use of EDX110 reduces the number of antibiotic treatments provided during the 16-week treatment period to the participant.
Systemic antibiotic usage in the full 24-week study period | 24 Weeks
  Determine if the use of EDX110 reduces the number of antibiotic treatments provided during the 24-week treatment period to the participant.
Incidence of new infections or increasing severity of infections during the 24-week study period | 24 Weeks
  Determine if the use of EDX110 reduces the number of infections in the index ulcer throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Mastandrea, MS, Study Director — ConvaTec Inc.
Locations (4):
- United States (4):
  - Axentra Bio, Phoenix, Arizona
  - Clemente Clinical Research, Santa Ana, California
  - ILD Research Center, Vista, California
  - Futuro Clinical Trials, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No